CLINICAL TRIAL: NCT05378451
Title: Totally Extraperitoneal Repair of Groin Hernia in Liver Transplanted Patients: a Case Series Study. (TOHER)
Brief Title: Totally Extraperitoneal Repair of Groin Hernia in Liver Transplanted Patients
Acronym: TOHER
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: TOHER2021
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2022-05

CONDITIONS: Liver Transplant Disorder; Liver Cirrhosis; Groin Hernia
Keywords: Liver Trasplant; Groin Hernia; Totally Extraperitoneal Repair
MeSH Terms: conditions — Liver Cirrhosis; Hernia, Inguinal | interventions — tetraethylpyrazine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Totally Extraperitoneal Groin Hernia Repair — Patients will undergo totally extraperitoneal groin hernia repair, by a single senior experimented surgeon and without modifications from the routine clinical practice due to study inclusion. TEP approach will be assessed by placement of 3 trocars in the lower midline. Preperitoneal space will be dissected under direct vision using Spacemaker Dissection Balloon (Applied Medical®). Systematic complete dissection of the myopectineal orifice, Retzius and Bogros spaces will be performed to identify all potential sites of hernia formation. It will be used a laparoscopic self-fixating mesh (ProGrip™). Preperitoneal instillation of local anesthesia (15 mL of 0.5% bupivacaine) will be placed placed by the surgeon under direct visualization into "triangle of pain". Local anesthesia (levobupivacaine 10mL 1%) will be applied in all the incisions.
  Other Names: TEP

SUMMARY:
Liver transplant recipients share the risk with cirrhotic patients for the development of inguinal hernias, but their liver failure pathophysiology has reversed following transplantation. Despite immunosuppression alters wound healing and infections, inguinal hernia repair in transplanted patients has shown better outcome compared to cirrhotic patients. Endoscopic inguinal hernia techniques have proved to be superior to open repair, due to lower incidence of postoperative complications and short-term convalescence, but there is no evidence of the use of this approach in liver transplanted patients. This prospective consecutive case series study will be the first study to describe the postoperative results of groin hernia repair in ambulatory surgery regimen in liver transplanted patients using totally extraperitoneal approach. The included patients will be prospectively registered in a standardized database. Rate of completion of surgery by totally extraperitoneal approach without the needing of conversion to anterior open approach or transabdominal preperitoneal approach due technical difficulties will be evaluated. Postoperative complications all along with quality standards criteria of ambulatory surgery will be reported for descriptive purposes.

DETAILED DESCRIPTION:
This will be a single center prospective consecutive case series study. Liver transplanted patients diagnosed of groin hernia will be operated using endoscopic totally extraperitoneal approach in ambulatory surgery regimen. Main objective will be to evaluate the rate of completion of surgery by totally extraperitoneal approach without the needing of conversion to anterior open approach or transabdominal preperitoneal approach due technical difficulties. Secondary objectives will be to record postoperative complications all along with quality standards criteria of ambulatory surgery.

The sample size could not be formally calculated as this is a pilot study. It is the first time that the surgical team has considered this type of surgical approach and we wish to evaluate the feasibility of this technique. Since in our center the number of surgical procedures of groin hernia in liver transplanted patients could be around 20 per year, for this pilot study we propose recruiting between 15-20 patients. The results will be representative of this type of surgical activities in a tertiary university hospital.

Liver transplanted patients diagnosed with groin hernia planned to undergo ambulatory surgical repair will be considered for being included in the study after informed consent. Perioperative management will be provided as determined by the local clinical practice without modifications due to study inclusion.The included patients will be prospectively registered in a standardized database. Background information and details regarding the surgery will be retrieved from the patients' medical records.

Information regarding postoperative complications will be collected up to 30 days after surgery. Following routine clinical practice, including telephonic contact on first postoperative 24h, clinical control follow up at 10 days and at month after the surgery.

This case series has been reported in line with the PROCESS Guideline.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age.
* Liver transplanted patients diagnosed from groin hernia and proposed for ambulatory surgery.
* Signed informed consent for inclusion in the study

Exclusion Criteria:

* Patients under 18 years of age.
* Pregnancy or breastfeeding.
* Inability to give informed consent.
* Patients not candidates for surgical treatment.
* Contraindication to general anesthesia.
* Procedures performed in an emergency setting.
* Patients non tributary to ambulatory surgery due to anesthesia management (ASA>III or decompensation in the last 3 months)
* Impossibility for the care of a responsible adult during first 24 hours after surgery.
* Domicile at a distance of more than 1 hour by vehicle from the hospital.
* Previous posterior approach for hernia repair.
* Previous cystectomy and prostatectomy surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Liver transplanted patients diagnosed with groin hernia planned to undergo ambulatory surgical repair will be considered for being included in the study after informed consent. Perioperative management will be provided as determined by the local clinical practice without modifications due to study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-05-08 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Rate of completion of surgery by totally extraperitoneal approach | 0 days (intraoperative)
  Rate of completion of surgery by totally extraperitoneal approach without the needing of conversion to anterior open approach or transabdominal preperitoneal approach due technical difficulties.

SECONDARY OUTCOMES:
Rate of intraoperative complications | 0 days (intraoperative)
  Register intraoperative complications (intestinal lesions, urinary bladder lesions, major vascular lesions...)
Rate of postoperative complications | 30 days (postoperative)
  Register postoperative complications (acute urinary retention, urinary infection, hematoma, seroma, surgical wound infection...)
Pain measurement | 10 days (postoperative).
  Control of pain assessed by Visual Analogue Score (at time of discharge, first postoperative day and after 10 days of surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Paula Dominguez-Garijo, MD, Principal Investigator — General Surgery, ICMDM, Hospital Clínic de Barcelona.
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR